CLINICAL TRIAL: NCT03224468
Title: Effect of Medical Marijuana on Neurocognition and Escalation of Use
Acronym: MMNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jodi Gilman, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015P001600
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-02

CONDITIONS: Pain; Insomnia; Depression; Anxiety
Keywords: medical marijuana; cannabis; pain; insomnia; depression; anxiety; addiction; dependence; neurocognition; MRI
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders; Marijuana Abuse; Behavior, Addictive | interventions — Medical Marijuana; nabiximols

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Marijuana Arm (Active Comparator): This group can begin using medical marijuana immediately.
  Interventions: Drug: Medical Marijuana
- Waitlist Control Arm (No Intervention): This group agrees to wait 3 months before using medical marijuana.

INTERVENTIONS:
Drug: Medical Marijuana — Patients in this group can choose when, where, and how much medical marijuana to use.
  Other Names: Cannabis
  Arms: Medical Marijuana Arm

SUMMARY:
This study will use a randomized controlled design to test whether patients who use medical marijuana, compared to a waitlist control group, experience a change in health outcomes (relief of symptoms, or adverse health outcomes such as new-onset symptoms of cannabis use disorders, neurocognitive impairments) or brain-based changes.

DETAILED DESCRIPTION:
This trial is a randomized, longitudinal study of medical marijuana (MM) that will: (1) characterize the impact of MM on indices of addiction, such as CUD, escalation of use, tolerance, and withdrawal among those who stop using, (2) assess, via dosing diaries, the effect of MM use patterns on use of other medications, and perception of underlying disease symptomatology, (3) characterize the impact of MM on neurocognitive performance, including executive function, memory, attention, and decision-making and (4) examine evidence for impact of MM on brain structure and function. This study will enroll 200 adults with no prior history of CUD or heavy marijuana use, who express interest in using MM to treat pain, insomnia, anxiety, and/or depression. Participants will be randomly assigned to either an active MM arm (n = 100), or to a waitlist control arm (WLC) (n = 100). Participants will be assessed at baseline, regularly for 3 months, and at a 6-month and 12-month follow-up for MM use behaviors, development of CUD, perception of disease symptomatology, and neurocognitive performance. Urine collected at each visit will be assessed with quantitative assays. MRI scans will be collected to longitudinally investigate possible brain changes associated with MM use.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-65 years, inclusive;
2. Competent and willing to provide written informed consent;
3. Desire to use medical marijuana for self-reported pain, sleep, or affective (mood and/or anxiety including PTSD) symptoms.
4. Not in possession of a medical marijuana card, but expressing intent to get one.
5. Able to communicate in English language.

Exclusion Criteria:

1. Current daily marijuana use (prior to enrollment)
2. Current substance use disorders (e.g. cocaine, opiate, stimulant). Light to moderate alcohol use is permitted (defined as 16 or less on the AUDIT), and nicotine dependence is permitted because of the high co-use of nicotine and marijuana. Participants cannot meet current SCID criteria for a use disorder on any illicit substance other than nicotine.
3. Pregnant (verified by a urine test).
4. In the opinion of the investigator, not able to safely participate in this study because of any medical or psychological issues (e.g. psychosis) that might compromise their safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 269 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jodi M Gilman, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Burdinski D, Kodibagkar A, Potter K, Schuster R, Evins AE, Ghosh S, Gilman J. Impact of year-long cannabis use for medical symptoms on brain activation during cognitive processes. medRxiv [Preprint]. 2024 May 1:2024.04.29.24306516. doi: 10.1101/2024.04.29.24306516. PMID 38746368
- [Derived] Livne O, Potter KW, Schuster RM, Gilman JM. Longitudinal Associations Between Cannabis Use and Cognitive Impairment in a Clinical Sample of Middle-Aged Adults Using Cannabis for Medical Symptoms. Cannabis Cannabinoid Res. 2024 Jun;9(3):e933-e938. doi: 10.1089/can.2022.0310. Epub 2023 Aug 25. PMID 37625034
- [Derived] Weiss JH, Tervo-Clemmens B, Potter KW, Evins AE, Gilman JM. The Cannabis Effects Expectancy Questionnaire-Medical (CEEQ-M): Preliminary psychometric properties and longitudinal validation within a clinical trial. Psychol Assess. 2023 Aug;35(8):659-673. doi: 10.1037/pas0001244. Epub 2023 Jun 8. PMID 37289502
- [Derived] Gilman JM, Potter K, Schuster RM, Hoeppner BB, Evins AE. Cannabis use for medical symptoms: Patterns over the first year of use. Addict Behav. 2023 Sep;144:107719. doi: 10.1016/j.addbeh.2023.107719. Epub 2023 Apr 13. PMID 37068366
- [Derived] Tervo-Clemmens B, Schmitt W, Wheeler G, Cooke ME, Schuster RM, Hickey S, Pachas GN, Evins AE, Gilman JM. Cannabis use and sleep quality in daily life: An electronic daily diary study of adults starting cannabis for health concerns. Drug Alcohol Depend. 2023 Feb 1;243:109760. doi: 10.1016/j.drugalcdep.2022.109760. Epub 2022 Dec 29. PMID 36638745
- [Derived] Gilman JM, Schuster RM, Potter KW, Schmitt W, Wheeler G, Pachas GN, Hickey S, Cooke ME, Dechert A, Plummer R, Tervo-Clemmens B, Schoenfeld DA, Evins AE. Effect of Medical Marijuana Card Ownership on Pain, Insomnia, and Affective Disorder Symptoms in Adults: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e222106. doi: 10.1001/jamanetworkopen.2022.2106. PMID 35302633

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Started | 173 | 96
Completed | 105 | 81
Not Completed | 68 | 15
Not completed — Did not obtain MM card | 53 | 0
Not completed — Lost to Follow-up | 4 | 11
Not completed — Cannabis Use Disorder at Baseline | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm | Total
Number analyzed (Participants) | 105 | 81 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (14.3) | 36.3 (14.5) | 37.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 50 | 122
  Male | 33 | 31 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 101 | 74 | 175
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 88 | 64 | 152
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 105 | 81 | 186
Education Level [Count of Participants; unit: Participants]
  High School | 4 | 6 | 10
  Part College | 16 | 20 | 36
  College 2 Years | 4 | 0 | 4
  College 4 Years | 35 | 26 | 61
  Part Grad School | 46 | 27 | 73
  Unknown | 0 | 2 | 2
Education Years [Mean (Standard Deviation); unit: years] | 16.6 (2.3) | 16.3 (2.7) | 16.5 (2.5)
Cannabis Use Frequency [Count of Participants; unit: Participants]
  Used less than weekly | 82 | 52 | 134
  Used weekly or more | 23 | 29 | 52
Primary Complaint [Count of Participants; unit: Participants]
  Pain | 37 | 24 | 61
  Insomnia | 22 | 20 | 42
  Anxiety/Depression | 46 | 37 | 83

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Number of Cannabis Use Disorder Symptoms Averaged Over 2, 4, and 12 Weeks
Description: The DSM-5 Cannabis Use Disorder (CUD) Checklist will evaluate symptoms of CUD (number of symptoms). The scale ranges from 0-11, with a higher score indicating a greater number of cannabis use disorder symptoms. A trained member of study staff assessed number of CUD symptoms through a structured interview. Each item was scored as "1" if the participant endorsed the symptom, and scored as "0" if they did not endorse the symptom. Reported results are an average taken over weeks 2, 4, and 12 to be consistent with the regression model estimates.
Time Frame: 2 weeks, 4 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 105 | 81
score on a scale | 0.39 (0.78) | 0.12 (0.48)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; The mean difference in number of symptoms between the MM and WLC groups was estimated via a linear model with a dummy-coded contrast (0 for WLC, 1 for MM). The model adjusted for change at weeks 4 and 12 of the study, and for a subject's number of symptoms at baseline; Test type: Superiority — Power was determined to be 85.2% using a Monte Carlo simulation approach in which data were simulated from a multi-level linear regression model with a subject-varying random intercept, a shared baseline across WLC and MMC, and fixed effects for a change over each time point. Simulated data were fit with a linear model estimated via GEE - simulations were repeated 1000 times and power was estimated as the proportion where the contrast between WLC and MM had p<0.05; p < 0.001, Regression, Linear — The p-value is adjusted for multiple comparisons using per Benjamini & Hochberg (1995) across the five primary outcome measures. Effects were deemed significant for p<0.05; Estimates were obtained using generalized estimating equations (GEE) with robust standard errors obtained by the sandwich estimator; Mean Difference (Net) = 0.28, 95% CI 2-sided [0.15 to 0.40], Standard Error of Mean 0.06 — Estimate is the mean difference in number of symptoms for MM above and beyond WLC (positive values denote higher number of symptoms for MM)

2. Primary Outcome: Mean Difference in Depression Subscale Scores From the HADS Averaged Over 2, 4, and 12 Weeks
Description: For those with depression symptoms, the depression subscale of the Hospital Anxiety and Depression Scale (HADS) will be used to assess symptoms. The subscale ranges from 0-21, with a higher score indicating worse depression outcomes. Reported results are an average taken over weeks 2, 4, and 12 to be consistent with the regression model estimates.
Time Frame: 2 weeks, 4 weeks, and 12 weeks
Population: The analysis is restricted to the subset of 83 participants out of 186 total who intended to use medical marijuana to address concerns for anxiety and depression.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 46 | 37
score on a scale | 5.4 (4.3) | 5.0 (3.9)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; The mean difference in scale scores between the MM and WLC groups was estimated via a linear model with a dummy-coded contrast (0 for WLC, 1 for MM). The model adjusted for change at weeks 4 and 12 of the study, and for a subject's scale scores at baseline; Test type: Superiority — Power was determined to be 83.6% using a Monte Carlo simulation approach in which data were simulated from a multi-level linear regression model with a subject-varying random intercept, a shared baseline across WLC and MMC, and fixed effects for a change over each time point. Simulated data were fit with a linear model estimated via GEE - simulations were repeated 1000 times and power was estimated as the proportion where the contrast between WLC and MM had p<0.05; p = 0.50, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.4 to 0.4], Standard Error of Mean 0.45 — Estimate is the mean difference in scale score for MM above and beyond WLC (positive values denote higher score for MM)

3. Primary Outcome: Mean Difference in Anxiety Subscale Scores From the HADS Averaged Over 2, 4, and 12 Weeks
Description: For those with anxiety symptoms, the anxiety subscale from the Hospital Anxiety and Depression Scale (HADS) will be used to assess symptoms. This subscale ranges from 0-21, with higher scores indicating worse anxiety outcomes. Reported results are an average taken over weeks 2, 4, and 12 to be consistent with the regression model estimates.
Time Frame: 2 Weeks, 4 Weeks, and 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 46 | 37
units on a scale | 8.4 (4.4) | 8.4 (3.8)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Power was determined to be 84.3% using a Monte Carlo simulation approach in which data were simulated from a multi-level linear regression model with a subject-varying random intercept, a shared baseline across WLC and MMC, and fixed effects for a change over each time point. Simulated data were fit with a linear model estimated via GEE - simulations were repeated 1000 times and power was estimated as the proportion where the contrast between WLC and MM had p<0.05; p = 0.90, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.30 to 0.24], Standard Error of Mean 0.5 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Mean Difference in Pain Severity Scores on the BPI Average Over 2, 4, and 12 Weeks
Description: For those with pain, the Brief Pain Inventory (BPI) severity subscale was used to assess pain symptoms. This scale ranges from 0-10, with a higher score indicating greater pain severity. Reported results are an average taken over weeks 2, 4, and 12 to be consistent with the regression model estimates.
Time Frame: 2 weeks, 4 weeks, and 12 weeks
Population: The analysis is restricted to the subset of 61 participants out of 186 total who intended to use medical marijuana to address concerns for pain.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 37 | 24
score on a scale | 2.7 (2.3) | 3.3 (2.5)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.93, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.38 to 0.39], Standard Error of Mean 0.5 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Mean Difference in Sleep Scores on the AIS Averaged Over 2, 4, and 12 Weeks
Description: For those with insomnia, the Athens Insomnia Scale (AIS) will be used to assess insomnia symptoms. This scale ranges from 0-24, with higher scores indicating worse sleep outcomes. Reported results are an average taken over weeks 2, 4, and 12 to be consistent with the regression model estimates.
Time Frame: 2 weeks, 4 weeks, and 12 weeks
Population: The analysis is restricted to the subset of 42 participants out of 186 total who intended to use medical marijuana to address concerns for insomnia.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 22 | 20
score on a scale | 8.8 (4.7) | 11.6 (3.7)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Power was determined to be 90.4% using a Monte Carlo simulation approach in which data were simulated from a multi-level linear regression model with a subject-varying random intercept, a shared baseline across WLC and MMC, and fixed effects for a change over each time point. Simulated data were fit with a linear model estimated via GEE - simulations were repeated 1000 times and power was estimated as the proportion where the contrast between WLC and MM had p<0.05; p < 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.79, 95% CI 2-sided [-1.30 to -0.43], Standard Error of Mean 0.7 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Mean Difference in Physical Health Scores on the SF-12 Averaged Over 2, 4, and 12 Weeks
Description: The Short Form-12 Health Survey (SF-12) Physical Health Summary Scale was used to assess self-report of physical health. SF-12 scores are based on an Item Response Theory model, in which they are z-scores rescaled to have a mean of 50 (SD=10) in any typical population. There are no range limits to this measure. Higher scores indicate better physical health functioning. Reported results are an average taken over weeks 2, 4, and 12 to be consistent with the regression model estimates.
Time Frame: 2 weeks, 4 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 105 | 81
score on a scale | 47.1 (11.0) | 48.2 (11.8)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; The mean difference in number of symptoms between the MM and WLC groups was estimated via a linear model with a dummy-coded contrast (0 for WLC, 1 for MM). The model adjusted for change at weeks 4 and 12 of the study, and for a subject's score at baseline; Test type: Superiority; Mean Difference (Net) = 0.8, 95% CI 2-sided [-1.0 to 2.5], Standard Error of Mean 0.9 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Mean Difference in Mental Health Scores on the SF-12 Averaged Over 2, 4, and 12 Weeks
Description: The Short Form 12 Health Survey (SF-12) Mental Health Summary Scale was used to assess self-report of mental health. SF-12 scores are based on an Item Response Theory model, in which they are z-scores rescaled to have a mean of 50 (SD=10) in any typical population. This measure has no range limits. Higher scores indicate better mental health functioning. Reported results are an average taken over weeks 2, 4, and 12 to be consistent with the regression model estimates.
Time Frame: 2 weeks, 4 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 105 | 81
score on a scale | 44.9 (11.7) | 41.5 (12.3)

8. Secondary Outcome: Mean Difference in Attention Switching Task: Congruency Cost Scores on the CANTAB Averaged Over 4 and 12 Weeks
Description: Congruency cost was assessed wth the Attention Switching Task (AST), which assesses attention shifting and executive function via a simple task assessing the direction (pointing left or right) and position (on the left or right side) of an arrow, and is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The range of this measure is -1900 to 1900 ms. It is calculated as the difference in the median latency for incongruent trials (i.e., trials where the direction of the arrow differs from the side it appears) minus the median latency for congruent trials (i.e., trials where the direction of the arrow matches the side it appears). Positive values indicate faster responses to congruent trials. Reported results are an average taken over weeks 4 and 12 to be consistent with the regression model estimates.
Time Frame: 4 weeks and 12 weeks
Population: The analysis is restricted to the subset of 162 participants out of 186 total who completed the AST module of the CANTAB at weeks 4 and 12.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 95 | 67
milliseconds (ms) | 63 (43) | 77 (50)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; The mean difference in number of symptoms between the MM and WLC groups was estimated via a linear model with a dummy-coded contrast (0 for WLC, 1 for MM). The model adjusted for change at week 12 of the study, and for a subject's score at baseline; Test type: Superiority; Mean Difference (Net) = -7.7, 95% CI 2-sided [-19.0 to 3.5], Standard Error of Mean 5.7 — Estimate is the mean difference in the congruency cost on response time for MM above and beyond WLC (positive values indicate higher cost for MM)

9. Secondary Outcome: Mean Difference in Attention Switching Task: Switching Cost Scores on the CANTAB Averaged Over 4 and 12 Weeks
Description: Switching cost was assessed with the Attention Switching Task (AST), which assesses attention shifting and executive function via a simple task assessing the direction (pointing left or right) and position (on the left or right side) of an arrow, and is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The range for this measure is -1900 to 1900 ms. It is calculated as the difference in the median latency for blocks of switching trials (i.e., blocks of trials where the response rule switches between indicating the direction of the arrow or the position of the arrow) minus the median latency for blocks of non-switching trials (i.e., blocks of trials where the response rule is always either to indicate the direction of the arrow or the position of the arrow across all trials). Positive scores indicate faster responses to non-switching trials. Reported results are an average taken over weeks 4 and 12 to be consistent with the regression model estimates.
Time Frame: 4 weeks and 12 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 95 | 67
milliseconds (ms) | 139 (90) | 162 (107)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = -24.1, 95% CI 2-sided [-45.9 to -2.2], Standard Error of Mean 11.2 — Estimate is the mean difference in the switching cost on response time for MM above and beyond WLC (positive values indicate higher cost for MM)

10. Secondary Outcome: Mean Difference in Rapid Visual Information Processing (RVP) Task: Discriminability Scores on the CANTAB Averaged Over 4 and 12 Weeks
Description: Discriminability was assessed with the Rapid Visual Information Processing (RVP) Task, which assesses sustained attention and is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). Discriminability scores are based on a transformation of response times and accuracy using the EZ-Diffusion model. There are no limits for this measure. Higher scores indicate that subjects can better discriminator between targets and distractors. Reported results are an average taken over weeks 4 and 12 to be consistent with the regression model estimates.
Time Frame: 4 weeks and 12 weeks
Population: The analysis is restricted to the subset of 177 participants out of 186 total who completed the RVP module of the CANTAB at weeks 4 and 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 101 | 76
score on a scale | 0.076 (0.047) | 0.058 (0.044)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.002, 95% CI 2-sided [-0.007 to 0.011], Standard Error of Mean 0.005 — Estimate is the mean difference in discriminability for MM above and beyond WLC (positive values indicate better ability to identify target items for MM)

11. Secondary Outcome: Mean Difference in Paired Associates Learning (PAL) Task: Total Errors Scores on the CANTAB Averaged Over 4 and 12 Weeks
Description: Total errors were assessed with the Paired Associates Learning (PAL) task, which assesses visual memory and is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The range for this measure is 0 to 70 errors. Higher scores indicate that the subject committed more errors (worse performance). Reported results are an average taken over weeks 4 and 12 to be consistent with the regression model estimates.
Time Frame: 4 weeks and 12 weeks
Population: The analysis is restricted to the subset of 177 participants out of 186 total who completed the PAL module of the CANTAB at weeks 4 and 12.
Measure: Mean (Standard Deviation); unit: Number of errors
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 101 | 76
Number of errors | 9.1 (11.3) | 9.3 (11.6)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.8 to 1.7], Standard Error of Mean 0.9 — Estimate is the mean difference in number of total errors for MM above and beyond WLC (positive values indicate greater number of errors for MM)

12. Secondary Outcome: Mean Difference in Spatial Working Memory (SWM) Task: Repetition Errors Scores on the CANTAB Averaged Over 4 and 12 Weeks
Description: Repetition errors were assessed with the Spatial Working Memory (SWM) task, which assesses spatial working memory and executive function. It is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The range for this measure is 0 to 63 errors. Higher scores indicate that more repetition errors were committed (worse performance). Reported results are an average taken over weeks 4 and 12 to be consistent with the regression model estimates.
Time Frame: 4 weeks and 12 weeks
Population: The analysis is restricted to the subset of 177 participants out of 186 total who completed the ? module of the CANTAB at weeks 4 and 12.
Measure: Mean (Standard Deviation); unit: Number of errors
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 101 | 76
Number of errors | 26.4 (18.4) | 30.0 (19.8)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = -3.6, 95% CI 2-sided [-7.4 to 0.3], Standard Error of Mean 2.0 — Estimate is the mean difference in number of repetition errors for MM above and beyond WLC (positive values indicate greater number of errors for MM)

13. Secondary Outcome: Mean Difference in Verbal Recognition Memory (VRM) Task: d' Scores on the CANTAB Averaged Over 4 and 12 Weeks
Description: Discriminability was assessed with the Verbal Recognition Memory task (VRM), which assess verbal memory. It is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). Discriminability scores are based on a transformation of hit and false alarm rates using a signal detection theory (SDT) model.There are no limits for this measure. Higher scores indicate that a subject was able to better discriminate between previously studied and novel words. Reported results are an average taken over weeks 4 and 12 to be consistent with the regression model estimates.
Time Frame: 4 weeks and 12 weeks
Population: The analysis is restricted to the subset of 171 participants out of 186 total who completed the VRM module of the CANTAB at weeks 4 and 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 98 | 73
score on a scale | 2.6 (0.8) | 2.7 (0.7)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.1 — Estimate is the mean difference in discriminability for MM above and beyond WLC (positive values indicate a greater ability to recognize previously studied words for MM)

14. Secondary Outcome: Mean Difference in Verbal Recognition Memory (VRM) Task: Free Recall Memory Scores on the CANTAB Averaged Over 4 and 12 Weeks
Description: Free Recall Memory was assessed with the Verbal Recognition Memory task (VRM), which assesses verbal memory. It is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The range for this measure is 0 to 18 words recalled. Higher scores indicate that subjects were able to correctly recall more previously studied words. Reported results are an average taken over weeks 4 and 12 to be consistent with the regression model estimates.
Time Frame: 4 weeks and 12 weeks
Population: The analysis is restricted to the subset of 175 participants out of 186 total who completed the free recall VRM module of the CANTAB at weeks 4 and 12.
Measure: Mean (Standard Deviation); unit: Total recalled
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
Number analyzed (Participants) | 101 | 74
Total recalled | 8.9 (2.7) | 8.5 (2.8)
Statistical Analysis 1: Comparison: Medical Marijuana Arm vs Waitlist Control Arm; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.2 to 1.0], Standard Error of Mean 0.3 — Estimate is the mean difference in number recalled for MM above and beyond WLC (positive values indicate a greater ability to recall previously studied words for MM)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 3 months.
Description: Adverse events are reported for baseline-3 months, as the primary outcomes were assessed at 3 months.
Arm/Group | Medical Marijuana Arm | Waitlist Control Arm
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/81
Serious Adverse Events (participants affected / at risk) | 1/105 | 0/81
Other Adverse Events (participants affected / at risk) | 90/105 | 60/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Marijuana Arm (N=105) | Waitlist Control Arm (N=81)
Cardiac Ablation (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Marijuana Arm (N=105) | Waitlist Control Arm (N=81)
Infections and infestations (Infections and infestations) | 50 | 31
Psychiatric symptoms (Psychiatric disorders) | 31 | 21
General disorders and conditions (General disorders) | 32 | 13
Nervous system symptoms (Nervous system disorders) | 13 | 8
Injury and poisoning (Injury, poisoning and procedural complications) | 12 | 10
Gastrointestinal disorders (Gastrointestinal disorders) | 14 | 5
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 2 | 8
Immune system disorders (Immune system disorders) | 4 | 5

LIMITATIONS AND CAVEATS:
Participants used variety of commercial medical cannabis products of their choice, at self-titrated doses; We do not attempt to comment on pharmacologic effects, risks, or benefits, of specific cannabinoids at specific doses; Inclusion based on self-reported symptoms, which may limit generalizability to those with formal diagnoses; Homogenous sample in terms of race, ethnicity; high dropout in the MMC group between randomization and baseline, reflecting cost and burden of obtaining a MMC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT03224468/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT03224468/ICF_001.pdf